CLINICAL TRIAL: NCT04512820
Title: Embryoscopic Evacuation of Early Missed Abortion Using the TRUCLEAR Hysteroscopic Morcellator System a Feasibility Study
Brief Title: Treatment of Missed Miscarriage With TRUCLEAR Tissue Removal System, a Feasiblity Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005-20-AAA
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2020-01

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TRUCLEAR TREATMENT (Experimental): patients up to 10 weeks of gestation with missed miscarriage undergoing evacuation of products of conception using the TRUCLEAR tissue removal system under direct hysteroscopic visualization
  Interventions: Device: TRUCLEAR tissue removal system

INTERVENTIONS:
Device: TRUCLEAR tissue removal system — evacuation of POC using the TRUCLEAR tissue removal system
  Other Names: non

SUMMARY:
the Aim of this study is to prospectively study the feasibility of evacuation of products of conception (POC) in missed miscarriages up to 10 weeks using the TRUCLEAR tissue removal system in order to achieve targeted treatment under direct vision of the POC and thus potentially reducing the risk of complications and intrauterine adhesions

DETAILED DESCRIPTION:
Embryoscopy and fetoscopy had been used increasingly in the treatment of missed abortions in the last two decades. This is done simply by transcervical hysteroscopy during pregnancy. The fact that we can directly view the embryo in the gestational sack allows us to document and describe the fetal morphology and to note different anatomical malformations. Phillips et al. described in 2001 the use of embryoscopy prior to evacuation of the uterus in early missed abortions in order to diagnose anatomical malformations and to allow sampling of the fetal tissues for genetic testing. This group also demonstrated that patients with repeated pregnancy loss are more likely to have morphologically normal embryos and less aneuploidy in cytogenetic analysis. The use of fetal tissue obtained in embryoscopy allows for more accurate genetic testing and diagnosis and reduces the number of maternal cells in the specimen.

Hysteroscopic morcellation had been used for intrauterine tissue extraction for over 20 years. Hysteroscopic morcellators have been shown to allow for rapid and complete resection of polyps, fibroids, uterine septa, and retained products of conception. These instruments use a rotating blade and a suction system that allows for the removal of the specimen under direct hysteroscopic visualization. When compared with standard resectoscopic technique, the use of hysteroscopic morcellators probably saves time and allows for more complete removal of the specimen.

Use of the hysteroscopic morcellator for resection of the fetal tissue in early missed abortions might prove beneficial over the standard blind Dilatation and curettage currently used to treat this condition. This technique might allow selective targeting of the fetal tissue thus decreasing the damage caused by trauma to the entire uterine cavity. In a recent systematic review the rate of intrauterine adhesions following D&C for missed abortions ranged between 16 to 21 percent. This technique was assessed in one case for a woman with previous Ashreman's syndrome and was found to be feasible although the authors state that visibility was poor while resecting the implantation site due to high vascularization.

The primary aim of the current study is to assess the feasibility of embryolysis - resection of an early missed abortion with the Truclear 8 mm hysteroscopic morcellator.

Secondary aims include the rate of complications, incomplete removal and intrauterine adhesions.

In this pilot feasibility study, we hypothesize that the 8mm Truclear Morcellator system will be able to achieve full evacuation of the uterine cavity. Performed under direct visualization and focused only on the implantation site, thus reducing the potential for further intrauterine adhesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with missed miscarriage up to 10 weeks from the last menstrual period
* Patients are able to provide written consent
* Patients with no underlying medical conditions

Exclusion Criteria:

* Inability to consent due to cognitive or language barrier
* Any underlying medical condition requiring medical treatment
* Documented failed hysteroscopy prior to the current referral
* Inability to consent due to cognitive or language barrier
* Uterine malformations or fibroids
* Previous cesarean section

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Number of cases with retained products of conception following the procedure | immediate - during the procedure
  Number of cases in which the procedure could not be completed using under vision hysteroscopic morcellation

SECONDARY OUTCOMES:
number of complications according to Dindo-Clavien scale | within six weeks from the procedure
  number of any complications according to the Dindo-Clavien scale, especially uterine perforation, infection, bleeding and pain that requires admission
incomplete removal | within 8 weeks
  number of patients with retained products of conception on ultrasound scan or hysteroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Ashdod University Hospital, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: Undecided
only unidentified data will be shared

REFERENCES:
- [Background] Philipp T, Kalousek DK. Transcervical embryoscopy in missed abortion. J Assist Reprod Genet. 2001 May;18(5):285-90. doi: 10.1023/a:1016666301481. PMID 11464580
- [Background] Feichtinger M, Wallner E, Hartmann B, Reiner A, Philipp T. Transcervical embryoscopic and cytogenetic findings reveal distinctive differences in primary and secondary recurrent pregnancy loss. Fertil Steril. 2017 Jan;107(1):144-149. doi: 10.1016/j.fertnstert.2016.09.037. Epub 2016 Oct 12. PMID 27743696
- [Background] Campos-Galindo I, Garcia-Herrero S, Martinez-Conejero JA, Ferro J, Simon C, Rubio C. Molecular analysis of products of conception obtained by hysteroembryoscopy from infertile couples. J Assist Reprod Genet. 2015 May;32(5):839-48. doi: 10.1007/s10815-015-0460-z. Epub 2015 Mar 17. PMID 25779005
- [Background] Shazly SA, Laughlin-Tommaso SK, Breitkopf DM, Hopkins MR, Burnett TL, Green IC, Farrell AM, Murad MH, Famuyide AO. Hysteroscopic Morcellation Versus Resection for the Treatment of Uterine Cavitary Lesions: A Systematic Review and Meta-analysis. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):867-77. doi: 10.1016/j.jmig.2016.04.013. Epub 2016 May 7. PMID 27164165
- [Background] Hooker A, Fraenk D, Brolmann H, Huirne J. Prevalence of intrauterine adhesions after termination of pregnancy: a systematic review. Eur J Contracept Reprod Health Care. 2016 Aug;21(4):329-35. doi: 10.1080/13625187.2016.1199795. PMID 27436757
- [Background] Harpham M, Abbott J. Use of a hysteroscopic morcellator to resect miscarriage in a woman with recurrent Asherman's syndrome. J Minim Invasive Gynecol. 2014 Nov-Dec;21(6):1118-20. doi: 10.1016/j.jmig.2014.05.006. Epub 2014 May 24. PMID 24865632
- [Derived] Weinberg S, Pansky M, Burshtein I, Beller U, Goldstein H, Barel O. A Pilot Study of Guided Conservative Hysteroscopic Evacuation of Early Miscarriage. J Minim Invasive Gynecol. 2021 Nov;28(11):1860-1867. doi: 10.1016/j.jmig.2021.04.017. Epub 2021 May 2. PMID 33951488